CLINICAL TRIAL: NCT06891287
Title: A Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of RT-114 in Healthy Volunteers
Brief Title: An Early Phase Study of RT-114
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RANI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT-114-001
Record Dates: First submitted 2025-03-07; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A is open label and Part B is randomized, double blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group A1 - Subcutaneous injection control (Active Comparator)
  Interventions: Drug: PG-102
- Group A2 - RT-114 (Experimental)
  Interventions: Combination Product: RT-114 is the RaniPill capsule with PG-102 for the treatment of obesity
- Group B1 - Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Group B2 - RT-114 (Experimental)
  Interventions: Combination Product: RT-114 is the RaniPill capsule with PG-102 for the treatment of obesity

INTERVENTIONS:
Combination Product: RT-114 is the RaniPill capsule with PG-102 for the treatment of obesity — RT-114 is the RaniPill capsule with PG-102 for the treatment of obesity.
  Arms: Group A2 - RT-114; Group B2 - RT-114
Drug: PG-102 — PG-102 is a drug for the treatment of obesity.
  Arms: Group A1 - Subcutaneous injection control
Other: Placebo — The placebo is the RaniPill with saline instead of a drug.
  Arms: Group B1 - Placebo

SUMMARY:
The goal of this Phase 1 study is to evaluate the safety and tolerability of RT-114 in healthy volunteers. The main objectives are:

Primary: To evaluate safety and tolerability of RT-114 when administered as single and multiple doses by assessing treatment emergent adverse events (TEAEs) in healthy volunteers

Secondary:

* To determine the pharmacokinetics of RT-114 administered as single and multiple doses
* To determine the pharmacodynamic effects of RT-114 administered as multiple doses

In the single dose portion of the study participants will either receive the drug via a subcutaneous injection or an oral pill (RT-114). In the repeat dose portion of the study participants will randomized to either RT-114 or a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ambulatory and between 18 to 65 years of age
2. Body mass index between:

   1. Part A: 19 - 32 kg/m2
   2. Part B: >30 kg/m2
3. Female volunteers must be non-pregnant or non-lactating during study participation
4. Male volunteers must agree to use acceptable forms of contraception, if necessary, and to not donate sperm during study participation
5. Have suitable venous access for blood sampling
6. In good general health confirmed by medical history, physical examination, and absence of clinically important laboratory abnormalities per Investigator's judgment
7. Participant understands the nature of the study, is willing to comply with protocol defined evaluations, and provide written informed consent

Exclusion Criteria:

1. History of intolerance to study drug (i.e., allergy to PG-102 or excipients).
2. HbA1c ≥ 6.5% at screening.
3. Treated with GLP-1 or GLP-2 agonist, or similar drugs, within 90 days prior to screening.
4. History of surgical treatment for obesity within 2 years (example: bariatric surgery, gastric banding, etc.) or gastrointestinal procedures for weight loss (including LAP-BAND®).
5. Total cholesterol >10.3 mmol/L or triglycerides ≥5.7 mmol/L (500 mg/dL) at screening.
6. Experienced a >5% loss in body weight within 2 months prior to screening.
7. History (≤10 years) or presence of disease determined by the PI to be clinically significant including:

   1. gastrointestinal/digestive (including diverticulitis, gastroparesis, stomach ulcers, inflammatory intestinal disease, gastrointestinal perforations/fistulae/intra-abdominal abscess, abnormal or irregular bowel movements)
   2. any other internal, non-gastrointestinal fistulae that is at an increased risk of bleeding
   3. hematological (including pancytopenia, aplastic anemia, or blood dyscrasia)
   4. proliferative retinopathy or maculopathy
   5. allergic disease excluding mild asymptomatic seasonal and food allergies
   6. renal, endocrine, hepatic, pulmonary (childhood asthma is allowed), neurologic, psychiatric, metabolic (including known diabetes mellitus)
8. Have a history of prolonged immunosuppressant therapy or photochemotherapy treatment.
9. Have a history of and/or current cardiac disease defined as one of the following:

   1. History of congestive heart failure; angina pectoris requiring anti-anginal medication.
   2. History of transmural infarction on ECG, if ECG results are available.
   3. History of sustained hypertension (systolic > 180 mmHg and/or diastolic > 100 mmHg), hypertensive crisis or hypertension encephalopathy.
   4. Clinically significant valvular heart disease, severe arterial thromboembolic events, or venous thromboembolic events.
10. Have a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus, human immunodeficiency virus (HIV) or history of active, latent, or inadequately treated tuberculosis (TB) infection.
11. Positive serum pregnancy test for women of childbearing potential at the Screening visit or positive urine pregnancy test with confirmatory serum pregnancy test prior to dosing.
12. Females who are breastfeeding.
13. Have a history of cancer including lymphoma, leukemia, and skin cancer (volunteers with a maximum of 3 surgically resected basal cell carcinoma or squamous cell carcinoma are permitted).
14. Any current active infections, including localized infections, or any recent history (within 1 week prior to study drug administration) of active infections (including severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] based on a positive COVID-19 polymerase chain reaction [PCR] nasopharyngeal swab test), cough or fever, or a history of recurrent or chronic infections.
15. Have had major surgery within 30 days prior to screening or will have an operation between screening and the end of study visit, or have any unhealed wound, including wound dehiscence and wound healing complications requiring medical intervention.
16. Have received live vaccines during the past 4 weeks before Screening or have the intention to receive vaccination during the study period or within 13 weeks after dosing.
17. Have received a Bacillus Calmette-Guerin (BCG) vaccination within 1 year prior to dose administration or is planning to receive a BCG vaccination within 1 year following dose administration.
18. History of alcohol abuse (defined as more than 14 standard drinks per week or more than 4 standard drinks on > 3 days per week; where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], 30 mL spirit [40% Alc./Vol]) within 12 weeks prior to the screening visit.
19. Excessive smoking habit (more than 5 cigarettes/day).
20. Positive drug or alcohol test results. In the event the urinary drug test is positive, the test may be repeated once (at the discretion of the PI) to confirm eligibility.
21. Consumption of any food containing poppy seeds within 48 hours prior to screening and admission to the clinical center.
22. Donation of more than 500 mL of blood within 4 weeks prior to drug administration.
23. Any history of non-traumatic hemorrhage (i.e., any hemorrhage requiring medical intervention) or any condition which may increase bleeding risk including clotting disorders, thrombocytopenia (platelet count < 150,000 per μL) or an international normalized ratio higher than 1.5.
24. Impaired liver function as determined by a serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 1.5 x upper limit of normal (ULN). Participants with values between ULN and 1.5 x ULN may be included in the study if considered not clinically significant by the Investigator.
25. Treatment with non-topical medications (including over-the-counter [OTC] medications and herbal remedies such as St. John's Wort extract) within 7 days or 5 half-lives of the drug (whichever is longer) prior to CTM administration, with the exception of birth control medications, multivitamins, vitamin C, food supplements and a limited amount of acetaminophen (up to 2 g in 24 hours, but <1 g in 4 hours) or ibuprofen (<1.2 g per day), which may be used throughout the study.
26. Participants on a higher than the lowest approved therapeutic dose regimen of proton pump inhibitors (see Section 9.1.7 for details).
27. Participants on a H2 receptor antagonists (e.g., famotidine, cimetidine).
28. History of proteinuria (other than trace amounts i.e., +, ++/+++).
29. Other clinically relevant findings per physical or laboratory examination or symptoms of a clinically relevant illness 3 weeks prior to the dose of study drug.
30. Participation in a clinical study with an investigational product (IP) dosing within 60 days or 5 half-lives of that IP (if known), whichever is longer, prior to IP administration in the current study.
31. History which, in the Investigator's judgement, makes the participant ineligible or exposes the participant to unacceptable risks.
32. Low likelihood, in the Investigator's judgment, to complete the study as required per study plan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of RT-114 by assessing treatment emergent adverse events (TEAEs) | Single dose and 8 weeks of repeat dosing

SECONDARY OUTCOMES:
To determine the pharmacokinetics of RT-114 | Single dose and 8 weeks of repeat dosing
  Peak Plasma Concentration (Cmax)
To determine the pharmacokinetics of RT-114 | Single dose and 8 weeks of repeat dosing
  Area under the plasma concentration versus time curve (AUC)
To determine the pharmacokinetics of RT-114 | Single dose and 8 weeks of repeat dosing
  Time to peak drug concentration (Tmax)
To determine the pharmacodynamic effects of RT-114 | Single dose and 8 weeks of repeat dose
  Body weight
To determine the pharmacodynamic effects of RT-114 | Single dose and 8 weeks of repeat dose
  Body mass index (BMI)
To determine the pharmacodynamic effects of RT-114 | Single dose and 8 weeks of repeat dose
  Waist circumference measurement
To determine the pharmacodynamic effects of RT-114 | Single dose and 8 weeks of repeat dose
  Waist-hip ratio

IPD SHARING:
Plan to Share IPD: Undecided